CLINICAL TRIAL: NCT05709301
Title: Multicenter, Randomized, Double-blinded, Placebo-controlled Clinical Trial of Donepezil for the Treatment of Mild Cognitive Impairment in Parkinson's Disease
Brief Title: Randomized Clinical Trial of Donepezil for the Treatment of Mild Cognitive Impairment in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIBSP-DON-2022-43
Record Dates: First submitted 2023-01-11; First posted 2023-02-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
Keywords: Parkinson's Disease-Mild Cognitive Impairment (PD-MCI); Donepezil; Randomized Clinical Trial (RCT)
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donepezil (Experimental)
  Interventions: Drug: Donepezil Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil Hydrochloride — Donepezil 10mg once daily
  Arms: Donepezil
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Phase II, multi-centric, randomized, double-blinded, placebo-controlled, parallel design clinical trial to evaluate the safety, tolerability and efficacy of Donepezil in patients with Mild Cognitive Impairment in Parkinson's Disease (PD-MCI). A total of 120 patients with PD-MCI will be randomized to 12 months of oral Donepezil 10mg or matching placebo (1:1).

Primary and co-primary efficacy endpoints are cognitive and functional cognitive scales: PD-CRS and PD-CFRS. Secondary efficacy endpoints include: cognitive tests evaluating attention, executive functions, language, memory and visuospatial domain; mood, anxiety, and apathy scales; questionnaires to evaluate quality of life; and subjective impression scales. Serum Neurofilament light chain, genetic screening of GBA, ApoE and MAPT, and Magnetic Resonance Imaging will be performed in a subset of these patients.

The study will be conducted in 20 different centers around Spain. The Movement Disorders Unit of the Neurology Department at Sant Pau Hospital (Barcelona, Spain) will be the coordinating center.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80
* PD diagnosis according to MDS criteria
* Hoehn and Yahr stage I-III
* Persistent subjective cognitive complaints for at least 6 months
* MDS PD-MCI Level I and Level II criteria
* Persistent PD-MCI for at least 3 months
* Stable dopaminergic treatment for at least 1 month

Exclusion Criteria:

* PD dementia criteria
* Severe motor complications
* DBS or any brain condition that may be contributing to cognitive impairment
* Active psychosis, major hallucinations, HADS ≥11, active impulse control disorder, or other active severe behavioral disorders.
* Treatment under anticholinergics, cholinergic enhancers, or neuroleptics.
* History of symptomatic arterial hypotension.
* Hypersensitivity or intolerance to donepezil or any of the excipients
* Pregnancy
* Unstable medical or surgical condition
* Any other significant observation that, in the investigator's opinion, would contraindicate participation in the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease-Cognitive Rating Scale (PD-CRS) | 12 months
  Global cognition
Parkinson's Disease-Cognitive Functional Rating Scale (PD-CFRS) | 12 months
  Cognitive functional performance

SECONDARY OUTCOMES:
Trail Making Test A (TMT-A) | 12 months
  Attention
TMT-B | 12 months
  Executive functions
Boston Naming Test | 12 months
  Language
Free and cued selective reminding test | 12 months
  Memory
Rey-Osterrieth complex figure test (ROCF) | 12 months
  Visuospatial
Hospital Anxiety and Depression Scale | 12 months
  Depression and Anxiety
Starkstein Apathy scale | 12 months
  Apathy
Neuropsychiatric Inventory | 12 months
  Hallucinations
Schwab & England scale | 12 months
  Quality of life
Clinical Global Impressions-Severity of illness | 12 months
  Subjective clinical change
CGI-Global improvement | 12 months
  Subjective clinical change
Patient Global Impression of Change | 12 months
  Subjective clinical change
8-item Parkinson's Disease Questionnaire | 12 months
  Quality of life
Judgment of Line Orientation | 12 months
  Visuspatial
recall of ROCF | 12 months
  Memory
Category fluency | 12 months
  Language
Phonemic Fluency | 12 months
  Executive functions
direct Digit Span | 12 months
  Attention

IPD SHARING:
Plan to Share IPD: No